CLINICAL TRIAL: NCT00534339
Title: EasyBand GOAL Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn to further optimize the device. No patients were enrolled in the trial.
Sponsor: Allergan Medical (Industry)
Responsible Party: Allergan Medical, Allergan
Organization: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10042
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2010-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

INTERVENTIONS:
Device: Easyband (Telemetrically adjustable gastric banding device) — EasyBand

SUMMARY:
Safety, effectiveness, and performance of Allergan's EasyBand telemetrically adjustable gastric banding device for the treatment of morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 3 year history of morbid obesity with documented failure of conservative, non-surgical means of weight reduction within 1 year prior to the screening visit;
* BMI >/= 40 kg/m2, or BMI >/= 35 kg/m2 and </= 40 kg/m2 with one or more significant medical conditions related to obesity;
* Candidate for surgical weight loss intervention

Exclusion Criteria:

* Previous surgical treatment of obesity;
* Patient already implanted with a device sensitive to radiofrequency emissions (implantable pacemaker, implantable defibrillator, etc);
* Physical or emotional conditions that may prohibit surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Percent excess weight loss (%EWL) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Allergan Medical, Study Director — Allergan Medical
Locations (2):
- USA, California, United States
- Canada, Quebec, Canada